CLINICAL TRIAL: NCT06046014
Title: Determining the Feasibility of Expressive Writing for Body Image Distress and Anxiety Among Adolescent and Young Adult Cancer Survivors
Brief Title: Feasibility of Expressive Writing for Body Image Distress and Anxiety Among Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: American Society of Clinical Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2023.079; HUM00239179 (Other: University of Michigan)
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Cancer; Young Adult Cancer; Body Image
Keywords: expressive writing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Writing (EW) (Experimental): four- week, in- home, Body Image (BI)- focused EW intervention
  Interventions: Other: BI Focused writing
- Attention Control (Active Comparator): four- week control writing program
  Interventions: Other: Control

INTERVENTIONS:
Other: BI Focused writing — BI Focused writing program
  Arms: Expressive Writing (EW)
Other: Control — Attention Control Writing
  Arms: Attention Control

SUMMARY:
Each year, about 89,500 adolescents and young adults (AYAs; 15-39 years old) are diagnosed with cancer and up to 60% experience body image (BI) distress. BI is largely developed in adolescence and young adulthood and has implications for self-identity and quality of life. Cancer itself and its associated treatments precipitate changes to appearance as well as body sensation and function, all of which can alter BI and lead to increased anxiety. An in-home BI-focused expressive writing (EW) program offers a promising outlet for addressing BI distress and anxiety in a way that eliminates constraints of clinical time and specialist availability.

There are no recommended interventions to help AYA cancer survivors cope with BI distress. To address this knowledge gap, the objective of this this pilot randomized-controlled trial is to determine the feasibility of a four-week BI-focused EW intervention to decrease BI distress and anxiety among AYA cancer survivors with the hypothesis that this intervention will reduce BI distress and anxiety.

DETAILED DESCRIPTION:
Protocol was updated to make the previous secondary outcome measures now exploratory

ELIGIBILITY:
Inclusion Criteria:

* Age 15-39 years
* History of one or more cancer diagnoses with all treatment (surgery, chemotherapy, radiation) completed ≥ 3 months before enrollment)
* BIS ≥10 at time of screening
* Ability to provide consent or assent and parental consent if applicable.

Exclusion Criteria:

* Plan to receive surgery, radiation, chemotherapy (including biologic agents, immunotherapy, and other targeted agents) for cancer treatment during the study period (from baseline assessment through post-four-week assessments and interview). Participants may continue with surveillance (such as imaging or biopsies) during the study period.
* Initiation of new treatments for body image distress or anxiety (e.g., pharmacologic, psychotherapy) ≤8 weeks prior to study enrollment. Although, participants may continue psychosocial or pharmacological treatments for anxiety or body image distress if the treatment were initiated at least eight weeks prior to study enrollment, the dose has not changed, and they report clinically relevant body image distress.
* History of limb-altering surgery or amputation (surgical exclusions are based on the premise that significant appearance-altering surgeries may impact body image distress differently than other cancer therapies)
* Currently receiving end-of-life care

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of in-home Body Image (BI) -focused expressive writing (EW) intervention for post-treatment adolescent and young adult (AYA) cancer survivors with BI distress (recruitment) | 7 months
  percent of patients recruited within 6 months
Feasibility of in-home Body Image (BI) -focused expressive writing (EW) intervention for post-treatment adolescent and young adult (AYA) cancer survivors with BI distress (adherence) | 7 months
  percent of patients who complete the baseline and four week patient reported measures. 50% of participants complete 3 out of 4 (75%) of the at-home writing interventions.
Feasibility of in-home Body Image (BI) -focused expressive writing (EW) intervention for post-treatment adolescent and young adult (AYA) cancer survivors with BI distress (practicality) | 7 months
  75% of participants complete the baseline and four-week patient-reported measures

OTHER OUTCOMES:
Acceptability of Intervention | 7 months
  4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale and score is reported as a calculated mean with higher scores indicating greater acceptability (no cut-off scores for interpretation are yet available). We will report descriptive statistics for this measure (mean and standard deviation) to quantitatively characterize perceive acceptability of the expressive writing intervention.
Facilitators and barriers of the intervention | 7 Months
  Qualitative interviews will be transcribed by a professional HIPAA compliant transcription agency. The Study team will analyze interview data using inductive content analysis will read transcripts to derive codes, discuss labels to group codes into categories, and identify major themes and corresponding exemplar quotes.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Wytiaz, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers